CLINICAL TRIAL: NCT01621490
Title: An Exploratory Study of the Biologic Effects of Nivolumab and Ipilimumab Monotherapy and Nivolumab in Combination With Ipilimumab Treatment in Subjects With Advanced Melanoma (Unresectable or Metastatic)
Brief Title: PH 1 Biomarker Study of Nivolumab and Ipilimumab and Nivolumab in Combination With Ipilimumab in Advanced Melanoma
Acronym: PD-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CA209-038; 2012-001840-23 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Advanced Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1-Cohort 1 and 2: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously Every 2 weeks, Up to 2 years depending on response
  Interventions: Biological: Nivolumab
- Part 2-Arm A: Nivolumab + Ipilimumab (Experimental): Nivolumab 1 mg/kg combined with Ipilimumab 3 mg/kg solution intravenously and then Nivolumab 3 mg/kg solution intravenously as specified
  Interventions: Biological: Nivolumab; Drug: Ipilimumab
- Part 3-Arm A: Nivolumab + Ipilimumab (Experimental): Nivolumab 1 mg/kg combined with Ipilimumab 3 mg/kg solution intravenously and then Nivolumab 3 mg/kg solution intravenously as specified
  Interventions: Biological: Nivolumab; Drug: Ipilimumab
- Part 3-Arm B: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously as specified
  Interventions: Biological: Nivolumab
- Part 4-Arm D: Nivolumab + Ipilimumab (Experimental): Nivolumab 1 mg/kg combined with Ipilimumab 3 mg/kg solution intravenously and then Nivolumab 3 mg/kg solution intravenously as specified
  Interventions: Biological: Nivolumab; Drug: Ipilimumab
- Part 4-Arm E: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously as specified
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558 (MDX1106)
Drug: Ipilimumab
  Other Names: BMS734016; Yervoy
  Arms: Part 2-Arm A: Nivolumab + Ipilimumab; Part 3-Arm A: Nivolumab + Ipilimumab; Part 4-Arm D: Nivolumab + Ipilimumab

SUMMARY:
The purpose of this study is to evaluate pharmacodynamic changes of Nivolumab and Nivolumab in combination with Ipilimumab treatment on the biomarkers measured in the peripheral blood and tumor tissues of subjects with advanced melanoma (unresectable or advanced)

DETAILED DESCRIPTION:
Allocation:

Part 1 and 2: Single Arm study

Part 3 and 4: Randomized Controlled Trial

Intervention Model:

Part 1 and 2: Single group: Single arm study

Part 3 and 4: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study

Minimum Age:

Part 1: 18

Part 2, 3 and 4: 16

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Part 1:

Inclusion Criteria:

* Men and women >18 years
* Eastern Cooperative Oncology Group (ECOG) status = 0 to 1
* Subjects with unresectable Stage III or IV melanoma who are either refractory or intolerant to, or have refused standard therapy for treatment of metastatic melanoma
* Subject must have histologic or cytologic confirmation of advanced melanoma
* Subjects must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Subjects must have at least 1 tumor site that can be biopsied at acceptable clinical risk and must consent to pre- and post-treatment biopsies

Exclusion Criteria:

* Active or progressing brain metastases
* Other concomitant malignancies (with some exceptions per protocol)
* Active or history of autoimmune disease
* Positive test for human immunodeficiency virus (HIV) 1&2 or known acquired immunodeficiency syndrome (AIDS)
* History of any hepatitis
* Prior therapy with any antibody/drug that targets the T cell coregulatory proteins, including but not limited to, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40,and anti-CD40 antibodies. However, half the patients must have progressed on anti Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA4) monoclonal antibody therapy

Part 2, 3 and 4:

Inclusion Criteria

* Men and women >16 years
* Eastern Cooperative Oncology Group (ECOG) status = 0 to 1
* Subjects with unresectable Stage III or IV melanoma who are either refractory or intolerant to, or have refused standard therapy for treatment of metastatic melanoma
* Subjects must never received anti-CTLA4 therapy
* Subjects must have histologic or cytologic confirmation of advanced melanoma
* Subjects must have at least two measurable lesions at baseline by CT or MRI as per RECIST 1.1 criteria
* Subjects must have at least 1 tumor site that can be biopsied at acceptable clinical risk and must consent to pre- and post-treatment biopsies
* Subjects in Part 4 must have brain metastases

Exclusion Criteria

* Active or progressing brain metastases (except for Part 4 subjects)
* Other concomitant malignancies (with some exceptions per protocol)
* Active or history of autoimmune disease
* Positive test for HIV 1&2 or known AIDS
* History of any hepatitis
* Prior therapy with any antibody/drug that targets the T cell coregulatory proteins, including but not limited to, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40,and anti-CD40 antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (12):
  - Ucla, Los Angeles, California
  - University Of Chicago, Chicago, Illinois
  - Sidney kimmel comprehensive cancer center at johns hopkins, Lutherville, Maryland
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
  - University Of Virginia, Charlottesville, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Local Institution - 0016, Amsterdam, Netherlands
- Local Institution - 0008, Pamplona, Spain

REFERENCES:
- [Derived] Kim YJ, Sheu KM, Tsoi J, Abril-Rodriguez G, Medina E, Grasso CS, Torrejon DY, Champhekar AS, Litchfield K, Swanton C, Speiser DE, Scumpia PO, Hoffmann A, Graeber TG, Puig-Saus C, Ribas A. Melanoma dedifferentiation induced by IFN-gamma epigenetic remodeling in response to anti-PD-1 therapy. J Clin Invest. 2021 Jun 15;131(12):e145859. doi: 10.1172/JCI145859. PMID 33914706
- [Derived] Anagnostou V, Bruhm DC, Niknafs N, White JR, Shao XM, Sidhom JW, Stein J, Tsai HL, Wang H, Belcaid Z, Murray J, Balan A, Ferreira L, Ross-Macdonald P, Wind-Rotolo M, Baras AS, Taube J, Karchin R, Scharpf RB, Grasso C, Ribas A, Pardoll DM, Topalian SL, Velculescu VE. Integrative Tumor and Immune Cell Multi-omic Analyses Predict Response to Immune Checkpoint Blockade in Melanoma. Cell Rep Med. 2020 Nov 17;1(8):100139. doi: 10.1016/j.xcrm.2020.100139. eCollection 2020 Nov 17. PMID 33294860
- [Derived] Stein JE, Soni A, Danilova L, Cottrell TR, Gajewski TF, Hodi FS, Bhatia S, Urba WJ, Sharfman WH, Wind-Rotolo M, Edwards R, Lipson EJ, Taube JM. Major pathologic response on biopsy (MPRbx) in patients with advanced melanoma treated with anti-PD-1: evidence for an early, on-therapy biomarker of response. Ann Oncol. 2019 Apr 1;30(4):589-596. doi: 10.1093/annonc/mdz019. PMID 30689736
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 170 participants were treated, 1 received ipilimumab monotherapy prior to the closure of Arm C in Amendment 06 and
  1 received an unplanned treatment; both were excluded from analysis. Analyses are presented for the remaining 168 treated participants.
Groups:
- N3 60 M Naive: Treatment Group: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; Naive = Anti-CTLA4 Naive
- N3 60M Prog: Treatment Group: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; PROG = Anti-CTLA4 Progressed
- N1 60M + I3 90M, W2: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion; W2 = Week 2 Biopsy
- N1 60M + I3 90M, W4: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion; W4 = Week 4 Biopsy
- N1 60M +I3 90M, WU: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion; WU = Unknown Week Biopsy
- N1 30M + I3 30M Non-BM; N1 30M +I3 30M BM: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 30M = 30 minute infusion; BM = Brain metastases
- N3 30M Non-BM: Treatment Group: N3 = Nivolumab 3mg/kg;30M = 30 minute infusion; BM = Brain metastases
- N3 30M BM: Treatment Group: N3 = Nivolumab 3mg/kg; 30M = 30 minute infusion; BM = Brain metastases
- I3 Monotherapy: Treatment Group: I3 = Ipilimumab 3 mg/kg infusion. Participant was enrolled prior to the closure of this arm via amendment
- Unplanned Treatment: Unplanned treatment of nivolumab 1 mg/kg x 4 then nivolumab 3 mg/kg
Period: Overall Study
Arm/Group | N3 60 M Naive | N3 60M Prog | N1 60M + I3 90M, W2 | N1 60M + I3 90M, W4 | N1 60M +I3 90M, WU | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M +I3 30M BM | N3 30M BM | I3 Monotherapy | Unplanned Treatment
Started | 41 | 44 | 11 | 10 | 6 | 25 | 11 | 10 | 10 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 41 | 44 | 11 | 10 | 6 | 24 | 11 | 10 | 10 | 1 | 1
Not completed — Subject no longer meets study criteria | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subject request to discontinue study | 1 | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse event unrelated to study drug | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Disease progression | 27 | 28 | 1 | 5 | 3 | 8 | 7 | 1 | 4 | 1 | 1
Not completed — Study drug toxicity | 1 | 4 | 5 | 3 | 1 | 10 | 1 | 4 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 7 | 6 | 4 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- N3 60M Prog: Treatment Group: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; PROG = Anti-CTLA4 Progressed;
- Total: Total of all reporting groups
Arm/Group | N3 60 M Naive | N3 60M Prog | N1 60M + I3 90M, W2 | N1 60M + I3 90M, W4 | N1 60M +I3 90M, WU | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M +I3 30M BM | N3 30M BM | I3 Monotherapy | Unplanned Treatment | Total
Number analyzed (Participants) | 41 | 44 | 11 | 10 | 6 | 25 | 11 | 10 | 10 | 1 | 1 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (12.49) | 53.7 (15.10) | 61.0 (11.82) | 58.5 (13.29) | 56.8 (9.64) | 56.9 (13.52) | 51.5 (15.55) | 56.9 (9.37) | 58.9 (13.46) | 52.0 (NA) — Standard deviation not calculated due to insufficient number of participants | 66.0 (NA) — Standard deviation not calculated due to insufficient number of participants | 55.9 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 3 | 4 | 3 | 8 | 4 | 4 | 5 | 1 | 0 | 69
  Male | 22 | 26 | 8 | 6 | 3 | 17 | 7 | 6 | 5 | 0 | 1 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 34 | 41 | 6 | 10 | 5 | 15 | 5 | 3 | 7 | 1 | 1 | 128
  Unknown or Not Reported | 5 | 3 | 3 | 0 | 1 | 10 | 5 | 6 | 3 | 0 | 0 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 41 | 43 | 11 | 10 | 6 | 25 | 11 | 10 | 10 | 1 | 1 | 169
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Change From Baseline to Week 7, of Interferon (IFN) and Interferon Gamma (IFN-gamma) Inducible Factors
Description: Baseline and post-treatment modulation of serum levels of chemokines, cytokines and other immune mediators were assessed by techniques that included ELISA or other multiplex-based assay methods. Primary analysis included IFN-gamma and IFN-gamma inducible factors, including chemokine [C-X-C motif] ligand 9 (CXCL9) and CXCL10
Time Frame: From last non-missing value prior to first dose to week 7 day 1
Population: All response evaluable participants who were treated per the protocol
Measure: Median (Standard Deviation); unit: pg/mL
Groups:
- N3 60M Naive: Treatment Group: Part 1: Nivolumab 3 mg/kg 60 Minute Infusion Anti-CTLA4 Naive
- N1 60M + I3 90M: Treatment Group: Part 2: Nivolumab 1 mg/kg 60 Minute Infusion + Ipilimumab 3 mg/kg 90 Minute
- N1 30M + I3 30M BM: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 30M = 30 minute infusion; BM = Brain metastases
- N1+ I3 Non-BM: Treatment Group: Part 2+3: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Non-Brain Metastases
- Naive Nivo Mono: Nivolumab Monotherapy CTLA-4 Naive
- All Nivo: Treatment Group: All Nivolumab Monotherapy
- All Combo: Treatment Group: All Combination Therapy
- Total: All treatments
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M + I3 30M BM | N3 30M BM | N1+ I3 Non-BM | Naive Nivo Mono | All Nivo | All Combo | Total
Number analyzed (Participants) | 40 | 40 | 27 | 23 | 11 | 8 | 7 | 50 | 58 | 98 | 58 | 156
pg/mL
  IFN-gamma Simoa: number analyzed (Participants) | 33 | 33 | 19 | 12 | 5 | 6 | 6 | 31 | 44 | 77 | 37 | 114
  IFN-gamma Simoa | 0.0130 (0.1740) | 0.0320 (0.0817) | 0.2310 (0.4528) | 0.1600 (1.2047) | 0.0520 (0.1207) | 0.0950 (1.5082) | 0.0375 (0.1868) | 0.2200 (0.8198) | 0.0130 (0.1674) | 0.0240 (0.1373) | 0.1520 (1.0023) | 0.0515 (0.5944)
  CXL9 (aka MIG): number analyzed (Participants) | 33 | 33 | 19 | 12 | 5 | 6 | 6 | 31 | 44 | 77 | 37 | 114
  CXL9 (aka MIG) | 1105.0 (10467.4) | 1890.0 (8706.0) | 4680.0 (18096.9) | 3542.0 (12133.1) | -29.0 (1684.2) | 5692.0 (6796.0) | 3610.0 (2197.4) | 458.5 (1651.0) | 1056.5 (9167.8) | 1235.0 (8984.2) | 4680.0 (14792.5) | 2027.0 (11491.9)
  CXL10 (aka IP10): number analyzed (Participants) | 33 | 33 | 19 | 12 | 5 | 6 | 6 | 31 | 44 | 77 | 37 | 114
  CXL10 (aka IP10) | 184.0 (514.1) | 160.0 (539.9) | 684.0 (2563.1) | 934.5 (2842.0) | 26.0 (172.7) | 514.0 (612.3) | 318.0 (354.0) | 695.0 (2627.7) | 185.0 (474.6) | 184.0 (500.7) | 684.0 (2450.6) | 234.5 (1566.3)

2. Primary Outcome: Tumor Infiltrating Lymphocytes (TILs) as Measured by Medians in Percent Positive CD8 and Positive CD4 at Baseline and On-treatment Biopsy, Both Using the Mosaic Singleplex IHC Assay
Description: Biomarkers examined were percent positive CD8 and percent positive CD4, both using the Mosaic Singleplex IHC assay. Analyses are presented with the medians at baseline and on-treatment, rather than the median change because the baseline values differed across groups. Baseline was defined as the last non-missing value on or prior to the first dose of study therapy. Biopsies were also collected on treatment.
Time Frame: From last non-missing value prior to first dose to week 4 day 1
Population: All response evaluable participants who were treated per the protocol
Measure: Median (Standard Deviation); unit: Percentage of positive cells
Groups:
- N1 60M + I3 90M W2: Treatment Group: Part 2: Nivolumab 1 mg/kg 60 Minute Infusion + Ipilimumab 3 mg/kg 90 Minute Infusion Week 2 Biopsy
- N1 60M + I3 90M W4: Treatment Group: Part 2: Nivolumab 1 mg/kg 60 Minute Infusion + Ipilimumab 3 mg/kg 90 Minute Infusion Week 4 Biopsy
- N3 30M + I3 30M BM: Treatment Group: Part 4: Nivolumab 1 mg/kg 30 Minute Infusion + Ipilimumab 3 mg/kg 30 Minute Infusion Brain Metastases
- Nivo Mono: Treatment Group: Part 1: Regular Infusion Nivolumab Mono
- Nivo Mono Reduced Infusion: Treatment Group: Reduced Infusion Nivolumab Monotherapy
- Week 2 Biopsy Combo: Treatment Group: Week 2 Biopsy Combo
- Week 2 Biopsy Non-BM Combo: Treatment Group: Week 2 Biopsy Non-Brain Metastases Combo
- Naive Nivo Mono Non-BM: Treatment Group: Naive Nivolumab Mono Non-Brain Metastases
- N1 + I3 Non-BM: Treatment Group: Part 2+3: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Non-Brain Metastases
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M W2 | N1 60M + I3 90M W4 | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N3 30M + I3 30M BM | N3 30M BM | Nivo Mono | Nivo Mono Reduced Infusion | Week 2 Biopsy Combo | Week 2 Biopsy Non-BM Combo | Naive Nivo Mono Non-BM | N1 + I3 Non-BM
Number analyzed (Participants) | 25 | 23 | 11 | 10 | 15 | 10 | 3 | 2 | 48 | 12 | 29 | 26 | 35 | 40
Percentage of positive cells
  Percent CD8 Baseline: number analyzed (Participants) | 21 | 21 | 11 | 10 | 15 | 10 | 3 | 2 | 42 | 12 | 29 | 26 | 31 | 40
  Percent CD8 Baseline | 3.730 (10.994) | 7.230 (10.712) | 3.260 (9.259) | 11.105 (9.524) | 4.700 (9.810) | 5.615 (12.475) | 18.590 (8.132) | 6.135 (5.664) | 6.360 (10.727) | 5.615 (11.472) | 4.700 (9.292) | 4.230 (9.401) | 5.210 (11.288) | 4.230 (9.844)
  Percent positive CD8 Week 2: number analyzed (Participants) | 0 | 0 | 10 | 0 | 8 | 9 | 3 | 2 | 0 | 11 | 21 | 18 | 9 | 18
  Percent positive CD8 Week 2 |  |  | 11.345 (21.316) |  | 7.970 (15.132) | 10.100 (10.909) | 8.470 (7.740) | 29.735 (5.254) |  | 10.910 (12.387) | 9.080 (17.510) | 9.125 (18.654) | 10.100 (10.909) | 9.125 (18.654)
  Percent positive CD8 Week 4: number analyzed (Participants) | 14 | 16 | 0 | 6 | 2 | 0 | 0 | 0 | 30 | 0 | 2 | 2 | 14 | 8
  Percent positive CD8 Week 4 | 18.435 (17.108) | 7.140 (25.204) |  | 32.455 (15.967) | 37.465 (5.706) |  |  |  | 15.150 (21.475) |  | 37.465 (5.706) | 37.465 (5.706) | 18.435 (17.108) | 34.785 (13.856)
  Percent CD4 Baseline: number analyzed (Participants) | 21 | 21 | 11 | 10 | 14 | 10 | 3 | 1 | 42 | 11 | 28 | 25 | 31 | 39
  Percent CD4 Baseline | 0.360 (1.844) | 0.600 (2.268) | 0.840 (1.852) | 0.470 (3.833) | 4.155 (6.624) | 4.950 (4.992) | 6.500 (8.108) | 2.780 (NA) — Standard deviation not calculated due to insufficient number of participants | 0.375 (2.057) | 4.600 (4.807) | 2.750 (5.833) | 2.610 (5.607) | 0.870 (3.727) | 1.510 (6.023)
  Percent positive CD4 Week 2: number analyzed (Participants) | 0 | 0 | 10 | 0 | 7 | 9 | 3 | 1 | 0 | 10 | 20 | 17 | 9 | 17
  Percent positive CD4 Week 2 |  |  | 4.500 (10.741) |  | 6.260 (8.518) | 4.210 (5.029) | 6.420 (14.778) | 20.830 (NA) — Standard deviation not calculated due to insufficient number of participants |  | 6.155 (6.585) | 6.125 (10.222) | 5.990 (9.602) | 4.210 (5.029) | 5.990 (9.602)
  Percent positive CD4 Week 4: number analyzed (Participants) | 14 | 16 | 0 | 6 | 2 | 0 | 0 | 0 | 30 | 0 | 2 | 2 | 14 | 8
  Percent positive CD4 Week 4 | 1.585 (3.071) | 1.260 (4.641) |  | 9.005 (13.324) | 24.520 (2.659) |  |  |  | 1.275 (3.921) |  | 24.520 (2.659) | 24.520 (2.659) | 1.585 (3.071) | 10.155 (12.707)

3. Secondary Outcome: Frequency of Adverse Events or Death
Description: The assessment of safety was based on frequency of deaths and adverse events (AEs). AEs were graded for severity according to the NCI CTCAE version 4.0.
Time Frame: Includes events reported between first dose and up to 100 days after last dose of study medication (up to approximately 73 months).
Population: All participants who received treatment per the protocol
Measure: Number; unit: Participants
Groups:
- N3 60M Naive: N3 = Nivolumab 3mg/kg;60M = 60 minute infusion; NAIVE = Anti-CTLA4 Naive
- N1 60M + I3 90M: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Participants
  Participants who died | 26 | 25 | 11 | 14 | 4 | 2 | 4
  Participants who died within 30 days of last dose | 3 | 2 | 4 | 0 | 0 | 1 | 0
  Participants who died within 100 days of last dose | 5 | 8 | 5 | 0 | 1 | 2 | 2
  Participants with an AE | 41 | 44 | 27 | 25 | 11 | 10 | 10

4. Secondary Outcome: Frequency of AEs Leading to Discontinuation of Study Drug and SAEs
Description: The assessment of safety was based on frequency of serious adverse events (SAEs) and adverse events (AEs) leading to discontinuation of study drug. AEs were graded for severity according to the NCI CTCAE version 4.0.
Time Frame: From enrollment to 100 days after the last dose date (up to approximately 73 months)
Population: All participants who received treatment per the protocol
Measure: Number; unit: Participants
Groups:
- N3 60M Naive: Part 1: Nivolumab 3 mg/kg 60 Minute Infusion Anti-CTLA4 Naive
- N3 60M Prog: Part 1: Nivolumab 3 mg/kg 60 Minute Infusion Anti-CTLA4 Progressed
- N1 60M + I3 90M: Part 2: Nivolumab 1 mg/kg 60 Minute Infusion + Ipilimumab 3 mg/kg 90 Minute Infusion
- N1 30M + I3 30M Non-BM: Part 3: Nivolumab 1 mg/kg 30 Minute Infusion + Ipilimumab 3 mg/kg 30 Minute Infusion Non-Brain Metastases
- N3 30M Non-BM: Part 3: Nivolumab 3 mg/kg 30 Minute Infusion Non-Brain Metastases
- N1 30M I3 30M BM: Part 4: Nivolumab 1 mg/kg 30 Minute Infusion + Ipilimumab 3 mg/kg 30 Minute Infusion Brain Metastases
Arm/Group | N3 60M Naive | N3 60M Prog | N1 60M + I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Participants
  SAEs | 20 | 22 | 20 | 14 | 2 | 7 | 4
  AEs Leading to Discontinuation | 2 | 6 | 12 | 9 | 1 | 4 | 2

5. Secondary Outcome: Number of Laboratory Abnormalities in Specific Liver Tests
Description: Abnormalities in hepatic parameters measured included those in aspartate aminotransferase (AST), alanine aminotransferase (ALT)and total bilirubin, with respect to upper limit of normal (ULN)
Time Frame: 101-120 days after last dose.
Population: Participants who were treated per the protocol and who had at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Number; unit: Events
Groups:
- N3 60M NAIVE: Treatment Group: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; Naive = Anti-CTLA4 Naive
- N1 60M +I3 90M: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion
Arm/Group | N3 60M NAIVE | N3 60M PROG | N1 60M +I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Events
  ALT OR AST > 3XULN: number analyzed (Participants) | 39 | 44 | 24 | 25 | 11 | 10 | 8
  ALT OR AST > 3XULN | 2 | 4 | 8 | 5 | 0 | 3 | 0
  ALT OR AST> 5XULN: number analyzed (Participants) | 39 | 44 | 24 | 25 | 11 | 10 | 8
  ALT OR AST> 5XULN | 1 | 2 | 6 | 4 | 0 | 1 | 0
  ALT OR AST> 10XULN: number analyzed (Participants) | 39 | 44 | 24 | 25 | 11 | 10 | 8
  ALT OR AST> 10XULN | 1 | 0 | 3 | 2 | 0 | 1 | 0
  ALT OR AST > 20XULN: number analyzed (Participants) | 39 | 44 | 24 | 25 | 11 | 10 | 8
  ALT OR AST > 20XULN | 0 | 0 | 1 | 0 | 0 | 1 | 0
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 39 | 44 | 25 | 24 | 11 | 10 | 8
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 2 | 1 | 0 | 2 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY: number analyzed (Participants) | 39 | 44 | 24 | 24 | 11 | 10 | 8
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 2 | 1 | 0 | 1 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAY: number analyzed (Participants) | 39 | 44 | 24 | 24 | 11 | 10 | 8
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAY | 0 | 0 | 2 | 1 | 0 | 1 | 0

6. Secondary Outcome: Number of Laboratory Abnormalities in Specific Thyroid Tests
Description: Abnormalities in thyroid parameters measured included those in thyroid stimulating hormone (TSH) levels with respect to upper limit of normal (ULN) and lower limit of normal (LLN)
Time Frame: 101-120 days after last dose.
Population: Participants who were treated per the protocol and who had at least one on-treatment measurement of TSH
Measure: Number; unit: Events
Arm/Group | N3 60M NAIVE | N3 60M PROG | N1 60M +I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 29 | 33 | 21 | 25 | 11 | 10 | 8
Events
  TSH > ULN | 9 | 16 | 7 | 7 | 1 | 3 | 4
  TSH > ULN WITH TSH <= ULN AT BASELINE | 4 | 9 | 7 | 4 | 1 | 3 | 2
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 0 | 0 | 3 | 3 | 0 | 2 | 2
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 9 | 16 | 4 | 4 | 1 | 1 | 2
  TSH < LLN | 3 | 4 | 11 | 12 | 2 | 6 | 5
  TSH <LLN WITH TSH >= LLN AT BASELINE | 3 | 4 | 11 | 12 | 2 | 6 | 5
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 0 | 5 | 4 | 0 | 2 | 2
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 0 | 3 | 1 | 0 | 0 | 1
  TSH < LLN WITH FT3/FT4 TEST MISSING | 3 | 4 | 3 | 7 | 2 | 4 | 2

7. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate (ORR) was defined as the percentage of participants with a best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized participants in the population of interest. The BOR was defined as the participant's best response designation, over the study as a whole, recorded between the date of first study drug administration and the date of objectively documented progression per RECIST 1.1, with subsequent confirmation, or date of subsequent anti-cancer therapy, whichever occurred first in the study.
Time Frame: Approximately every 8 weeks until disease progression and in follow-up if no progression (up to approximately 73 months)
Population: All participants who received treatment per the protocol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- N3 60M Prog: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion;PROG = Anti-CTLA4 Progressed;
- N1 60M+I3 90M: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion
- N1 30M + I3 30M BM: N3 = Nivolumab 3mg/kg; I3 = Ipilimumab 3 mg/kg; 30M = 30 minute infusion; BM = Brain metastases
Arm/Group | N3 60M Naive | N3 60M Prog | N1 60M+I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Percentage of participants | 31.7 [18.1 to 48.1] | 22.7 [11.5 to 37.8] | 44.4 [25.5 to 64.7] | 40.0 [21.1 to 61.3] | 27.3 [6.0 to 61.0] | 70.0 [34.8 to 93.3] | 60.0 [26.2 to 87.8]

8. Secondary Outcome: Median Duration of Response (mDOR)
Description: Median duration of response (mDOR) was calculated for subjects with BOR of CR or PR only, and is defined as time between the date of first documented objective response and the date of the first subsequent disease progression or death, whichever occurred first, if death occurred within 100 days after last dose of study medication.
Time Frame: From date of first documented objective response to date of disease progression or death, up to approximately 27 months
Population: All participants who received treatment per the protocol
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- N1 30M + I3 30M NON-BM: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 30M = 30 minute infusion; BM = Brain metastases
- N3 30M NON-BM: N3 = Nivolumab 3mg/kg; 30M = 30 minute infusion; BM = Brain metastases
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M NON-BM | N3 30M NON-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Months | 16.59 [7.29 to NA] — Upper limit not reached due to insufficient number of events | NA [5.55 to NA] — Median and upper limit not reached due to insufficient number of events | NA [5.85 to NA] — Median and upper limit not reached due to insufficient number of events | 26.25 [7.85 to NA] — Upper limit not reached due to insufficient number of events | NA [3.71 to NA] — Median and upper limit not reached due to insufficient number of events | NA [22.01 to NA] — Median and upper limit not reached due to insufficient number of events | 20.27 [13.57 to NA] — Upper limit not reached due to insufficient number of events

9. Secondary Outcome: Median Time to Response (mTTR)
Description: Median time to response (mTTR) for a participant with a BOR of CR or PR is defined as the time from the first dosing date to the date of the first documented objective response (CR or PR).
Time Frame: From the first dosing date to the date of the first documented objective response, up to approximately 15 months
Population: All participants who received treatment per the protocol
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M NON-BM | N3 30M NON-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Months | 1.87 [1.77 to 3.71] | 2.78 [1.84 to 14.59] | 1.41 [1.28 to 1.87] | 2.51 [1.28 to 2.86] | 1.41 [1.41 to 6.90] | 1.71 [1.38 to 7.43] | 2.14 [1.25 to 4.99]

10. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) for a participant was defined as the time from the date of first dose of study medication to the date of the first documented disease progression, or death due to any cause, whichever occurred first, if death occurred within 100 days after last dose of study medication.
Time Frame: From first dose of study medication to the date of progression or death, whichever occurs first, up to approximately 29 months
Population: All participants who received treatment per the protocol
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M NON-BM | N3 30M NON-BM | N1 30M + I3 30M BM | N3 30M BM
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10
Months | 3.68 [1.84 to 7.36] | 5.62 [1.87 to 9.66] | 7.00 [1.41 to NA] — Upper limit not reached due to insufficient number of events | 9.69 [1.94 to 29.01] | 4.93 [1.41 to NA] — Upper limit not reached due to insufficient number of events | NA [1.18 to NA] — Median and upper limit not reached due to insufficient number of events | 23.00 [0.85 to NA] — Upper limit not reached due to insufficient number of events

11. Secondary Outcome: Immunogenicity of Nivolumab and Nivolumab in Combination With Ipilimumab as Measured by the Number of Serum Anti-drug Antibody (ADA) Positive Participants and the Number of Neutralizing ADA Positive Participants
Description: Time Frame: Part 1: Day 1, Day 15, Day 43 of cycle 1, Day 1 of cycle 2, Day 15 of cycle 3, every 16 weeks after cycle 3 up to 2 years, follow-up visit 1 (40-60 days after last treatment), and follow-up visit 2 (101-120 days since last treatment) Part 2, 3 and 4: Weeks 1, 3, 4, 7, 9, 10, 13, 25, 53, 79, 95 follow-up visit 1 (40-60 days after last treatment), and follow-up visit 2 (101-120 days since last treatment)
Time Frame: Up to follow-up visit 2 (101-120 days since last treatment)
Population: A subset of all participants who were treated per the protocol who had a baseline and at least 1 post-baseline ADA assessment for nivolumab and ipilimumab separately
Measure: Number; unit: Participants
Groups:
- N1 60M + I3 (Nivo ADA; N1 60M + I3 90M (Ipi ADA): Part 2: Nivolumab 1 mg/kg 60 Minute Infusion + Ipilimumab 3 mg/kg 90 Minute
- N1 30M + I3 30M Non-BM (Nivo ADA); N1 30M + I3 30M Non-BM (Ipi ADA): Part 3: Nivolumab 1 mg/kg 30 Minute Infusion + Ipilimumab 3 mg/kg 30 Minute Infusion Non-Brain Metastases
- N1 30M + I3 30M (Nivo ADA); N1 30M + I3 30M (Ipi ADA): Part 4: Nivolumab 1 mg/kg 30 Minute Infusion + Ipilimumab 3 mg/kg 30 Minute Infusion Brain Metastases
- Total (Nivo ADA); Total (Ipi ADA): Total (All Nivolumab or Nivolumab + Ipilimumab Treated Subjects with Baseline and at Least One Post-Baseline Assessment)
Arm/Group | N3 60M NAIVE | N3 60M PROG | N1 60M + I3 (Nivo ADA | N1 60M + I3 90M (Ipi ADA) | N1 30M + I3 30M Non-BM (Nivo ADA) | N1 30M + I3 30M Non-BM (Ipi ADA) | N3 30M Non-BM | N1 30M + I3 30M (Nivo ADA) | N1 30M + I3 30M (Ipi ADA) | N3 30M BM | Total (Nivo ADA) | Total (Ipi ADA)
Number analyzed (Participants) | 38 | 42 | 22 | 22 | 24 | 23 | 11 | 10 | 9 | 7 | 154 | 54
Participants
  ADA positive | 2 | 5 | 10 | 1 | 16 | 4 | 1 | 7 | 0 | 1 | 42 | 5
  Neutralizing ADA positive: number analyzed (Participants) | 2 | 5 | 10 | 1 | 16 | 4 | 1 | 7 | 0 | 1 | 42 | 5
  Neutralizing ADA positive | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 |  | 0 | 3 | 0

12. Secondary Outcome: Objective Response Rate (ORR) by PD-L1 Expression
Description: For immunohistochemistry (IHC) measurements, to explore the PD-L1 expression as a potential predictive marker of clinical activity, PD-L1 expression status were derived from percent of tumor cells exhibiting cell surface staining for PD-L1 at baseline and/or in archived biopsy samples using verified and/or validated assays. In the case of multiple specimens, a subject would be identified as PD-L1 expression levels >= x%, where x% can be 10%, 5%, and/or 1% in any of the baseline and/or archived specimens. The association between PD-L1 expression status and/or level and clinical efficacy measures was assessed. The objective response rate (ORR) was defined as the number of subjects with a best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized subjects in the population of interest (all response-evaluable participants).
Time Frame: as for outcome 7
Population: All participants who received treatment per the protocol
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- N3 60M NAIVE, W4: Treatment Group: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; NAIVE = Anti-CTLA4 Naive
- N3 60M PROG, W4: Treatment Group: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; PROG = Anti-CTLA4 Progressed;
- N1 60M + I3 90M, WU: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 90M = 90 minute infusion; 60M = 60 minute infusion; WU = Unknown Week Biopsy
- N3 30M NON-BM, W2; N3 30M BM, W2; N3 30M, W2: Treatment Group: N3 = Nivolumab 3mg/kg; 30M = 30 minute infusion; W2 = Week 2 Biopsy
- N1 30M + I3 30M BM, W2: Treatment Group: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; 30M = 30 minute infusion; W2 = Week 2 Biopsy
- N3 60M, W4: N3 = Nivolumab 3mg/kg; 60M = 60 minute infusion; W4 = Week 4 Biopsy
- N1 + I3, W2: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; W2 = Week 2 Biopsy
- N1 + I3 W2, NON-BM: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; W2 = Week 2 Biopsy; BM = Brain metastases
- N3 NAIVE, NON-BM: N3 = Nivolumab 3mg/kg; NAIVE = Anti-CTLA4 Naive; BM = Brain metastases
- N1 + I3 NON-BM: N1 = Nivolumab 1mg/kg; I3 = Ipilimumab 3 mg/kg; BM = Brain metastases
Arm/Group | N3 60M NAIVE, W4 | N3 60M PROG, W4 | N1 60M + I3 90M, W2 | N1 60M + I3 90M, W4 | N1 60M + I3 90M, WU | N1 30M + I3 30M NON-BM | N3 30M NON-BM, W2 | N1 30M + I3 30M BM, W2 | N3 30M BM, W2 | N3 60M, W4 | N3 30M, W2 | N1 + I3, W2 | N1 + I3 W2, NON-BM | N3 NAIVE, NON-BM | N1 + I3 NON-BM | Total
Number analyzed (Participants) | 39 | 36 | 11 | 10 | 6 | 22 | 9 | 4 | 3 | 75 | 12 | 37 | 33 | 48 | 49 | 140
Percentage of Participants
  STTU 1 - 1% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 20 | 17 | 7 | 6 | 2 | 11 | 5 | 2 | 1 | 37 | 6 | 20 | 18 | 25 | 26 | 71
  STTU 1 - 1% Level PD-L1 Status: Met criteria | 40.0 [19.1 to 63.9] | 35.3 [14.2 to 61.7] | 85.7 [42.1 to 99.6] | 50.0 [11.8 to 88.2] | 50.0 [1.3 to 98.7] | 63.6 [30.8 to 89.1] | 40.0 [5.3 to 85.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 37.8 [22.5 to 55.2] | 50.0 [11.8 to 88.2] | 75.0 [50.9 to 91.3] | 72.2 [46.5 to 90.3] | 40.0 [21.1 to 61.3] | 65.4 [44.3 to 82.8] | 50.7 [38.6 to 62.8]
  STTU 1 - 5% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 10 | 9 | 5 | 5 | 1 | 7 | 2 | 2 | 1 | 19 | 3 | 14 | 12 | 12 | 18 | 42
  STTU 1 - 5% Level PD-L1 Status: Met criteria | 40.0 [12.2 to 73.8] | 33.3 [7.5 to 70.1] | 80.0 [28.4 to 99.5] | 60.0 [14.7 to 94.7] | 100.0 [2.5 to 100.0] | 71.4 [29.0 to 96.3] | 50.0 [1.3 to 98.7] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 36.8 [16.3 to 61.6] | 66.7 [9.4 to 99.2] | 78.6 [49.2 to 95.3] | 75.0 [42.8 to 94.5] | 41.7 [15.2 to 72.3] | 72.2 [46.5 to 90.3] | 57.1 [41.0 to 72.3]
  STTU 1 - 10% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 7 | 5 | 3 | 4 | 1 | 3 | 1 | 2 | 1 | 12 | 2 | 8 | 6 | 8 | 11 | 27
  STTU 1 - 10% Level PD-L1 Status: Met criteria | 42.9 [9.9 to 81.6] | 20.0 [0.5 to 71.6] | 100.0 [29.2 to 100.0] | 75.0 [19.4 to 99.4] | 100.0 [2.5 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 33.3 [9.9 to 65.1] | 100.0 [15.8 to 100.0] | 87.5 [47.3 to 99.7] | 83.3 [35.9 to 99.6] | 50.0 [15.7 to 84.3] | 81.8 [48.2 to 97.7] | 63.0 [42.4 to 80.6]

13. Secondary Outcome: Duration of Response (DOR) by PD-L1 Expression
Description: For immunohistochemistry (IHC) measurements, to explore the PD-L1 expression as a potential predictive marker of clinical activity, PD-L1 expression status were derived from percent of tumor cells exhibiting cell surface staining for PD-L1 at baseline and/or in archived biopsy samples using verified and/or validated assays. In the case of multiple specimens, a subject would be identified as PD-L1 expression levels >= x%, where x% can be 10%, 5%, and/or 1% in any of the baseline and/or archived specimens. Median duration of response (mDOR) was calculated for all response-evaluable participants with best overall response of CR or PR only, and is defined as time between the date of first documented objective response and the date of the first subsequent disease progression or death, whichever occurred first, if death occurred within 100 days after last dose of study medication.
Time Frame: From the date of first documented objective response and the date of the first subsequent disease progression or death, whichever occurred first, up to approximately 73 months
Population: All response evaluable participants who were treated per the protocol
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | N3 60M NAIVE, W4 | N3 60M PROG, W4 | N1 60M + I3 90M, W2 | N1 60M + I3 90M, W4 | N1 60M + I3 90M, WU | N1 30M + I3 30M NON-BM | N3 30M NON-BM, W2 | N1 30M + I3 30M BM, W2 | N3 30M BM, W2 | N3 60M, W4 | N3 30M, W2 | N1 + I3, W2 | N1 + I3 W2, NON-BM | N3 NAIVE, NON-BM | N1 + I3 NON-BM | Total
Number analyzed (Participants) | 39 | 36 | 11 | 10 | 6 | 22 | 9 | 4 | 3 | 75 | 12 | 37 | 33 | 48 | 49 | 140
Months
  STTU 1 - 1% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 20 | 17 | 7 | 6 | 2 | 11 | 5 | 2 | 1 | 37 | 6 | 20 | 18 | 25 | 26 | 71
  STTU 1 - 1% Level PD-L1 Status: Met criteria | 15.21 [4.60 to 18.20] | NA [15.57 to NA] — Median and upper limit not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limit not reached due to insufficient number of events. | NA [NA to NA] — Median, lower limit and upper limit not reached due to insufficient number of events. | NA [NA to NA] — Median, lower limit and upper limit not reached due to insufficient number of events. | 26.25 [8.31 to NA] — Upper limit not reached due to insufficient number of events. | NA [3.71 to NA] — Median and upper limit not reached due to insufficient number of events. | 22.01 [NA to NA] — Upper and lower limits not reached due to insufficient number of events. | NA [NA to NA] — Median, upper and lower limits not reached due to insufficient number of events. | 16.59 [11.50 to NA] — Upper limit not reached due to insufficient number of events. | NA [3.71 to NA] — Median and upper limit not reached due to insufficient number of events. | 26.25 [22.01 to NA] — Upper limit not reached due to insufficient number of events. | NA [8.31 to NA] — Median and upper limit not reached due to insufficient number of events. | 15.21 [3.71 to NA] — Upper limit not reached due to insufficient number of events. | NA [26.25 to NA] — Median and upper limit not reached due to insufficient number of events. | 26.25 [16.59 to NA] — Upper limit not reached due to insufficient number of events.
  STTU 1 - 5% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 10 | 9 | 5 | 5 | 1 | 7 | 2 | 2 | 1 | 19 | 3 | 14 | 12 | 12 | 18 | 42
  STTU 1 - 5% Level PD-L1 Status: Met criteria | 15.21 [11.50 to 16.59] | NA [15.57 to NA] — Median and upper limit not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limit not reached due to insufficient number of events. | NA [NA to NA] — Median, lower limit and upper limit not reached due to insufficient number of events. | NA [NA to NA] — Median, lower limit and upper limit not reached due to insufficient number of events. | 26.25 [8.31 to NA] — Upper limit not reached due to insufficient number of events. | NA [3.71 to NA] — Median and upper limits not reached due to insufficient number of events. | 22.01 [NA to NA] — Lower and upper limits not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | 16.59 [11.50 to NA] — Upper limit not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | 26.25 [8.31 to NA] — Upper limit not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limits not reached due to insufficient number of events. | 16.59 [11.50 to NA] — Upper limit not reached due to insufficient number of events. | NA [8.31 to NA] — Median and upper limits not reached due to insufficient number of events. | 26.25 [15.57 to NA] — Upper limit not reached due to insufficient number of events.
  STTU 1 - 10% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 7 | 5 | 3 | 4 | 1 | 3 | 1 | 2 | 1 | 12 | 2 | 8 | 6 | 8 | 11 | 27
  STTU 1 - 10% Level PD-L1 Status: Met criteria | 15.90 [15.21 to 16.59] | 15.57 [NA to NA] — Lower and upper limits not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limit not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | 22.01 [NA to NA] — Lower and upper limits not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | 15.57 [15.21 to 16.59] | NA [NA to NA] — Median, lower and upper limits not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limits not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limits not reached due to insufficient number of events. | 16.59 [15.21 to NA] — Upper limit not reached due to insufficient number of events. | NA [2.96 to NA] — Median and upper limits not reached due to insufficient number of events. | NA [15.57 to NA] — Median and upper limits not reached due to insufficient number of events.

14. Secondary Outcome: Progression Free Survival (PFS) by PD-L1 Expression
Description: For immunohistochemistry (IHC) measurements, to explore the PD-L1 expression as a potential predictive marker of clinical activity, PD-L1 expression status were derived from percent of tumor cells exhibiting cell surface staining for PD-L1 at baseline and/or in archived biopsy samples using verified and/or validated assays. In the case of multiple specimens, a subject would be identified as PD-L1 expression levels >= x%, where x% can be 10%, 5%, and/or 1% in any of the baseline and/or archived specimens. The association between PD-L1 expression status and/or level and clinical efficacy measures was assessed. The progression free survival rate (PFSR) for a subject was defined as the time from the date of first dose of study medication to the date of the first documented disease progression, or death due to any cause, whichever occurred first, if death occurred within 100 days after last dose of study medication.
Time Frame: as for outcome 10
Population: All response evaluable participants who were treated per the protocol
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | N3 60M NAIVE, W4 | N3 60M PROG, W4 | N1 60M + I3 90M, W2 | N1 60M + I3 90M, W4 | N1 60M + I3 90M, WU | N1 30M + I3 30M NON-BM | N3 30M NON-BM, W2 | N1 30M + I3 30M BM, W2 | N3 30M BM, W2 | N3 60M, W4 | N3 30M, W2 | N1 + I3, W2 | N1 + I3 W2, NON-BM | N3 NAIVE, NON-BM | N1 + I3 NON-BM | Total
Number analyzed (Participants) | 39 | 36 | 11 | 10 | 6 | 22 | 9 | 4 | 3 | 75 | 12 | 37 | 33 | 48 | 49 | 140
Months
  STTU 1 - 1% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 20 | 17 | 7 | 6 | 2 | 11 | 5 | 2 | 1 | 37 | 6 | 20 | 18 | 25 | 26 | 71
  STTU 1 - 1% Level PD-L1 Status: Met criteria | 4.50 [1.84 to 15.18] | 9.66 [3.71 to NA] — Upper limit not reached due to insufficient number of events | NA [1.22 to NA] — Median and upper limit not reached due to insufficient number of events | NA [0.85 to NA] — Median and upper limit not reached due to insufficient number of events | NA [0.76 to NA] — Median and upper limit not reached due to insufficient number of events | 29.01 [1.94 to 29.01] | 8.77 [1.22 to NA] — Upper limit not reached due to insufficient number of events | NA [23.95 to NA] — Median and upper limit not reached due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | 6.24 [3.65 to 17.05] | 8.77 [1.22 to NA] — Upper limit not reached due to insufficient number of events | 29.01 [4.17 to NA] — Upper limit not reached due to insufficient number of events | 29.01 [3.02 to NA] — Upper limit not reached due to insufficient number of events | 5.36 [1.94 to 10.94] | 29.01 [3.02 to NA] — Upper limit not reached due to insufficient number of events | 10.58 [5.62 to 19.81]
  STTU 1 - 5% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 10 | 9 | 5 | 5 | 1 | 7 | 2 | 2 | 1 | 19 | 3 | 14 | 12 | 12 | 18 | 42
  STTU 1 - 5% Level PD-L1 Status: Met criteria | 6.28 [0.33 to 17.05] | 19.29 [1.77 to NA] — Upper limit not reached due to insufficient number of events | NA [1.22 to NA] — Median and upper limit not reached due to insufficient number of events | NA [0.85 to NA] — Median and upper limit not reached due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | 29.01 [1.94 to 29.01] | NA [1.22 to NA] — Median and upper limit not reached due to insufficient number of events | NA [23.95 to NA] — Median and upper limit not reached due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | 7.20 [1.87 to 18.40] | NA [1.22 to NA] — Median and upper limit not reached due to insufficient number of events | 29.01 [3.02 to NA] — Upper limit not reached due to insufficient number of events | 29.01 [1.94 to NA] — Upper limit not reached due to insufficient number of events | 6.28 [1.22 to 17.05] | 29.01 [3.02 to NA] — Upper limit not reached due to insufficient number of events | 17.05 [5.36 to 29.01]
  STTU 1 - 10% Level PD-L1 Status: Met criteria: number analyzed (Participants) | 7 | 5 | 3 | 4 | 1 | 3 | 1 | 2 | 1 | 12 | 2 | 8 | 6 | 8 | 11 | 27
  STTU 1 - 10% Level PD-L1 Status: Met criteria | 5.36 [0.33 to 18.40] | 19.29 [1.77 to 19.29] | NA [4.17 to NA] — Median and upper limit not reached due to insufficient number of events | NA [1.64 to NA] — Median and upper limit not reached due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | NA [1.94 to NA] — Median and upper limit not reached due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | NA [23.95 to NA] — Median and upper limit not reached due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | 6.24 [1.71 to 18.40] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events | NA [1.94 to NA] — Median and upper limit not reached due to insufficient number of events | NA [1.94 to NA] — Median and upper limit not reached due to insufficient number of events | 11.20 [0.33 to NA] — Upper limit not reached due to insufficient number of events | NA [1.94 to NA] — Median and upper limit not reached due to insufficient number of events | 19.29 [5.36 to NA] — Upper limit not reached due to insufficient number of events

15. Secondary Outcome: Overall Survival Rate (OSR)
Description: The percentage of participants surviving to time t, where t is a specific length of time, eg, 12 months, which was determined by the available data for final analysis and was documented in the DPP. The percentage was calculated by the product-limit method (Kaplan-Meier estimate), which takes into account censored data. The overall survival rate (OSR) for a participant was defined as the time from the date of first dose of study medication to the date of death for any cause. A participant who had not died was censored at last known date alive.
Time Frame: From first dose of study medication to the date of death for any cause, up to approximately 73 months
Population: All participants who were treated per the protocol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- N3 NAIVE: N3 = Nivolumab 3mg/kg; NAIVE = Anti-CTLA4 Naive
- All N3: N3 = Nivolumab 3mg/kg
- N1 + I3: All combination
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M NON-BM | N3 30M NON-BM | N1 30M + I3 30M BM | N3 30M BM | N1 + I3 NON-BM | N3 NAIVE | All N3 | N1 + I3 | Total
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10 | 52 | 62 | 106 | 62 | 168
Percentage of participants
  3 months | 92.7 [79.0 to 97.6] | 90.8 [77.3 to 96.4] | 85.2 [65.2 to 94.2] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 90.0 [47.3 to 98.5] | 80.0 [40.9 to 94.6] | 92.3 [80.8 to 97.0] | 90.2 [79.6 to 95.5] | 90.5 [83.0 to 94.8] | 91.9 [81.7 to 96.6] | 91.0 [85.5 to 94.5]
  6 months | 85.3 [70.2 to 93.1] | 78.9 [63.3 to 88.4] | 81.5 [61.1 to 91.8] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 90.0 [47.3 to 98.5] | 80.0 [40.9 to 94.6] | 90.4 [78.4 to 95.9] | 85.3 [73.6 to 92.0] | 82.6 [73.8 to 88.6] | 90.3 [79.7 to 95.5] | 85.5 [79.2 to 90.1]
  9 months | 75.0 [58.5 to 85.7] | 71.7 [55.5 to 82.8] | 81.5 [61.1 to 91.8] | 88.0 [67.3 to 96.0] | 90.0 [47.3 to 98.5] | 90.0 [47.3 to 98.5] | 68.6 [30.5 to 88.7] | 84.6 [71.6 to 92.0] | 76.6 [63.7 to 85.4] | 74.6 [64.9 to 81.9] | 85.5 [74.0 to 92.2] | 78.7 [71.6 to 84.2]
  12 months | 72.4 [55.7 to 83.7] | 64.5 [48.2 to 76.9] | 77.6 [56.8 to 89.3] | 88.0 [67.3 to 96.0] | 80.0 [40.9 to 94.6] | 90.0 [47.3 to 98.5] | 68.6 [30.5 to 88.7] | 82.6 [69.3 to 90.6] | 73.1 [59.8 to 82.6] | 69.5 [59.5 to 77.5] | 83.8 [72.0 to 91.0] | 74.9 [67.5 to 80.9]
  24 months | 51.0 [34.3 to 65.4] | 46.8 [31.1 to 61.1] | 69.6 [48.3 to 83.5] | 58.1 [36.0 to 75.0] | 58.3 [23.0 to 82.1] | 80.0 [40.9 to 94.6] | 57.1 [21.7 to 81.5] | 64.3 [49.3 to 75.8] | 53.3 [39.6 to 65.2] | 50.6 [40.3 to 60.0] | 66.8 [53.3 to 77.2] | 56.8 [48.7 to 64.1]

16. Secondary Outcome: Percent Probability for Progression Free Survival Rate (PFSR)
Description: The Progression Free Survival Rate (PFSR) is defined as the probability of a participant remaining progression free or survival to time t, where t is equal to the specified timepoints. This probability will be calculated by the product limit method (Kaplan-Meier estimates) which takes into account censored data.
  Medians and 95% confidence interval are estimated using the Kaplan-Meier method. If there is an insufficient number of events, the median and confidence intervals cannot be calculated.
Time Frame: From first dose up to the specified timepoints of 3, 6, 9, 12, and 24 months
Population: All participants treated per the protocol
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | N3 60M Naive | N3 60M PROG | N1 60M + I3 90M | N1 30M + I3 30M Non-BM | N3 30M Non-BM | N1 30M + I3 30M BM | N3 30M BM | N1+ I3 Non-BM | Naive Nivo Mono | All Nivo | All Combo | Total
Number analyzed (Participants) | 41 | 44 | 27 | 25 | 11 | 10 | 10 | 52 | 62 | 106 | 62 | 168
Percent probability
  3 months | 53.7 [37.4 to 67.4] | 59.1 [43.2 to 71.9] | 54.6 [34.0 to 71.2] | 69.3 [46.1 to 84.0] | 54.5 [22.9 to 78.0] | 77.8 [36.5 to 93.9] | 70.0 [32.9 to 89.2] | 61.3 [46.2 to 73.3] | 56.5 [43.3 to 67.7] | 57.5 [47.6 to 66.3] | 63.6 [49.8 to 74.6] | 59.5 [51.5 to 66.6]
  6 months | 38.7 [24.0 to 53.2] | 47.1 [31.8 to 61.0] | 50.7 [30.6 to 67.7] | 60.1 [37.2 to 76.9] | NA [NA to NA] — The median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | 77.8 [36.5 to 93.9] | 70.0 [32.9 to 89.2] | 55.0 [40.0 to 67.6] | 44.3 [31.5 to 56.3] | 45.4 [35.6 to 54.7] | 58.2 [44.3 to 69.7] | 49.8 [41.8 to 57.3]
  9 months | 33.2 [19.3 to 47.8] | 42.2 [27.3 to 56.3] | 42.2 [23.2 to 60.2] | 55.0 [37.2 to 76.9] | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | 77.8 [36.5 to 93.9] | 70.0 [32.9 to 89.2] | 48.0 [33.2 to 61.3] | 38.5 [26.1 to 50.7] | 40.0 [30.4 to 49.4] | 52.3 [38.5 to 64.4] | 44.2 [36.3 to 51.8]
  12 months | 30.4 [17.0 to 45.0] | 34.3 [20.4 to 48.6] | 42.2 [23.2 to 60.2] | 36.7 [16.2 to 57.6] | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | 77.8 [36.5 to 93.9] | 70.0 [32.9 to 89.2] | 40.1 [25.8 to 54.0] | 34.7 [22.7 to 46.9] | 34.4 [25.2 to 43.8] | 45.8 [32.1 to 58.5] | 38.3 [30.6 to 46.0]
  24 months | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | 21.8 [10.2 to 36.2] | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | 40.1 [25.8 to 54.0] | NA [NA to NA] — Median, the lower limit, and the upper limit were not calculated because there was an insufficient number of events to calculate using the Kaplan-Meier method. | 18.2 [10.7 to 27.3] | 42.3 [28.2 to 55.7] | 26.5 [19.2 to 34.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 73 months). Serious Adverse events and other adverse events were assessed from date of first dose to 100 days following date of last dose (up to approximately 73 months).
Groups:
- N3 30M Non-BM; N3 30M BM: Treatment Group: N3 = Nivolumab 3mg/kg; 30M = 30 minute infusion; BM = Brain metastases
Arm/Group | N3 60M NAIVE | N3 60M PROG | N1 60M + I3 90M, W2 | N1 60M + I3 90M, W4 | N1 60M + I3 90M, WU | N1 30M + I3 30M Non-BM | N3 30M Non-BM | I3 Monotherapy | N1 30M + I3 30M BM | N3 30M BM | Unplanned Treatment
All-Cause Mortality (participants affected / at risk) | 26/41 | 25/44 | 4/11 | 3/10 | 4/6 | 14/25 | 4/11 | 1/1 | 2/10 | 4/10 | 1/1
Serious Adverse Events (participants affected / at risk) | 20/41 | 22/44 | 8/11 | 6/10 | 6/6 | 14/25 | 2/11 | 1/1 | 7/10 | 4/10 | 1/1
Other Adverse Events (participants affected / at risk) | 41/41 | 44/44 | 11/11 | 10/10 | 6/6 | 25/25 | 10/11 | 1/1 | 10/10 | 9/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N3 60M NAIVE (N=41) | N3 60M PROG (N=44) | N1 60M + I3 90M, W2 (N=11) | N1 60M + I3 90M, W4 (N=10) | N1 60M + I3 90M, WU (N=6) | N1 30M + I3 30M Non-BM (N=25) | N3 30M Non-BM (N=11) | I3 Monotherapy (N=1) | N1 30M + I3 30M BM (N=10) | N3 30M BM (N=10) | Unplanned Treatment (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8 | 0 | 2 | 3 | 4 | 1 | 0 | 1 | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arachnoiditis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N3 60M NAIVE (N=41) | N3 60M PROG (N=44) | N1 60M + I3 90M, W2 (N=11) | N1 60M + I3 90M, W4 (N=10) | N1 60M + I3 90M, WU (N=6) | N1 30M + I3 30M Non-BM (N=25) | N3 30M Non-BM (N=11) | I3 Monotherapy (N=1) | N1 30M + I3 30M BM (N=10) | N3 30M BM (N=10) | Unplanned Treatment (N=1)
Anaemia (Blood and lymphatic system disorders) | 9 | 8 | 0 | 2 | 2 | 5 | 0 | 1 | 2 | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 2 | 0 | 1 | 4 | 0 | 0 | 3 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 2 | 3 | 3 | 0 | 4 | 0 | 0 | 1 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 5 | 5 | 1 | 3 | 2 | 5 | 0 | 0 | 3 | 1 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vision blurred (Eye disorders) | 2 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 5 | 3 | 1 | 3 | 4 | 3 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 11 | 14 | 4 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 14 | 5 | 5 | 2 | 9 | 4 | 0 | 6 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 6 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 12 | 3 | 2 | 3 | 13 | 4 | 0 | 7 | 2 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4 | 2 | 2 | 2 | 9 | 1 | 0 | 3 | 1 | 1
Asthenia (General disorders) | 3 | 1 | 3 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Chills (General disorders) | 3 | 4 | 3 | 4 | 1 | 3 | 0 | 0 | 2 | 2 | 0
Fatigue (General disorders) | 21 | 29 | 7 | 4 | 4 | 13 | 5 | 1 | 6 | 6 | 1
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 4 | 3 | 2 | 1 | 1 | 3 | 1 | 0 | 3 | 3 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 9 | 6 | 1 | 3 | 2 | 6 | 0 | 0 | 4 | 1 | 0
Pain (General disorders) | 3 | 11 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 11 | 9 | 6 | 6 | 3 | 9 | 3 | 0 | 5 | 3 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 2 | 5 | 3 | 2 | 5 | 0 | 0 | 2 | 0 | 0
Amylase increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 2 | 6 | 3 | 2 | 6 | 0 | 0 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 4 | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Cortisol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 8 | 8 | 2 | 2 | 2 | 3 | 0 | 0 | 3 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Norovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 8 | 5 | 2 | 2 | 2 | 3 | 0 | 1 | 0 | 1 | 1
Weight increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 15 | 5 | 3 | 2 | 4 | 1 | 1 | 4 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 3 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 2 | 4 | 2 | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 13 | 2 | 3 | 2 | 5 | 1 | 0 | 3 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 8 | 1 | 1 | 2 | 1 | 3 | 0 | 2 | 2 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 10 | 9 | 0 | 3 | 3 | 9 | 0 | 0 | 5 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 5 | 1 | 3 | 2 | 2 | 1 | 0 | 3 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spermatic cord haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 4 | 3 | 2 | 4 | 1 | 0 | 3 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 3 | 3 | 3 | 5 | 1 | 0 | 2 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 12 | 8 | 3 | 2 | 8 | 1 | 0 | 4 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 11 | 11 | 5 | 3 | 1 | 6 | 1 | 0 | 1 | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 5 | 2 | 4 | 0 | 4 | 0 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 4 | 6 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 6 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased activity (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fine motor delay (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤ 60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT01621490/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT01621490/SAP_002.pdf